CLINICAL TRIAL: NCT00364299
Title: Prevention of Ventilator-Associated Pneumonia by Automatic Control of the Tracheal Tube Cuff Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other); Sociedad Española de Neumología y Cirugía Torácica (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FIS 020744
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Last update posted 2006-10-20 (Estimated); Status verified 2006-05

CONDITIONS: Ventilator-Associated Pneumonia; Mechanical Ventilation
Keywords: Ventilator-associated pneumonia; Mechanical ventilation; Tracheal tube cuff pressure
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

INTERVENTIONS:
Device: Automatic control of tracheal tube cuff pressure

SUMMARY:
Background: The aspiration of contaminated secretions pooled above the endotracheal tube cuff secondary to inadvertent falls of cuff pressure is the main pathogenic mechanism of ventilator-associated pneumonia (VAP). Aim of the study: To assess the efficacy of an automatic device for the continuous regulation of tracheal tube cuff pressure in decreasing the incidence of VAP.

DETAILED DESCRIPTION:
Design: Prospective, randomized, controlled trial, with 2 groups: study (automated control of cuff pressure) and control (standard control of cuff pressure). Setting: Respiratory Intensive Care Unit (RICU). Subjects: Patients >18 yr, intubated and ventilated. Interventions and measurements: Study group (cuff pressure will be kept constant at 25 cmH2O with the automatic device) and control group (cuff pressure control every 8 h. at the same level using a manual pressure controller, according with standard routine); recording of clinical variables at admission and during RICU stay, and end-point variables (incidence of VAP, etiologic microorganisms, RICU and hospital stay, RICU and 60-d mortality. Expected results: Lower incidence of VAP in study group, compared with control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years,
* Orotracheal intubation for less than 24 hours
* Expectancy to remain on mechanical ventilation for more than 48 hours

Exclusion Criteria:

* Pneumonia
* Witnessed macroscopic aspiration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142
Dates: Start 2002-10; Study Completion 2006-05

PRIMARY OUTCOMES:
Incidence of ventilator-associated pneumonia

CONTACTS AND LOCATIONS:
Overall Officials: Miquel Ferrer, MD, Principal Investigator — Hospital Clinic, Barcelona,Spain.
Locations (1):
- Servei de Pneumologia, Hospital Clinic, Barcelona, Barcelona, Spain